CLINICAL TRIAL: NCT02814695
Title: Can Yeast Cells Emulate Vitamin E on In-vitro Protection of Human Spermatozoa Against Oxidative Stress?
Brief Title: Yeast Cells as Antioxidant-Producing Probiotics
Acronym: Probiotics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Benha University (Other)
Collaborators: Hawaa Fertility Center (Other); Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed Saad, Assistant professor of Ob.&Gyn., Benha University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HAWAA-001
Record Dates: First submitted 2016-06-21; First posted 2016-06-28 (Estimated); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Infertility, Male
Keywords: Male infertility; oxidative stress; antioxidants; probiotics; Vitamin E; Baker's Yeast
MeSH Terms: conditions — Infertility, Male | interventions — Yeast, Dried

STUDY DESIGN:
Intervention Model Description: control, vit E, vit C, Yeast
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): First fraction was control, 0.1ml of liquefied semen mixed with 0.1ml Ham's F10 medium and incubated at 37o C for 30 minutes.
- Vit E supplementation (Experimental): 0.1ml liquefied semen was mixed with 0.1ml Ham's F10 medium supplemented with (2 mg/ml) Vitamin E and incubated at 37o C for 30 minutes.
  Interventions: Dietary Supplement: Vit E
- Yeast supplementation (Experimental): 0.1ml liquefied semen was mixed with 0.1ml Ham's F10 medium supplemented with (20 mg/ml) Yeast extraction and incubated at 37o C for 30 minutes.
  Interventions: Dietary Supplement: Yeast
- Vit C supplementation (Experimental): fractions (Vit. C. 1,2,3), 0.1ml liquefied semen was mixed with 0.1ml Ham's F10 medium supplemented with (0.02, 0.04, 0.06 mg/ml) Vitamin C respectively and incubated at 37o C for 30 minutes.
  Interventions: Dietary Supplement: Vit C 1; Dietary Supplement: Vit C 2; Dietary Supplement: Vit C 3

INTERVENTIONS:
Dietary Supplement: Vit E — 0.1ml liquefied semen was mixed with 0.1ml Ham's F10 medium supplemented with (2 mg/ml) Vitamin E and incubated at 37o C for 30 minutes.
  Arms: Vit E supplementation
Dietary Supplement: Yeast — 0.1ml liquefied semen was mixed with 0.1ml Ham's F10 medium supplemented with (20 mg/ml) yeast extraction and incubated at 37o C for 30 minutes.
  Arms: Yeast supplementation
Dietary Supplement: Vit C 1 — 0.1ml liquefied semen was mixed with 0.1ml Ham's F10 medium supplemented with (0.02 mg/ml) Vitamin C and incubated at 37o C for 30 minutes.
  Arms: Vit C supplementation
Dietary Supplement: Vit C 2 — 0.1ml liquefied semen was mixed with 0.1ml Ham's F10 medium supplemented with (0.04 mg/ml) Vitamin C and incubated at 37o C for 30 minutes.
  Arms: Vit C supplementation
Dietary Supplement: Vit C 3 — 0.1ml liquefied semen was mixed with 0.1ml Ham's F10 medium supplemented with (0.06 mg/ml) Vitamin C and incubated at 37o C for 30 minutes.
  Arms: Vit C supplementation

SUMMARY:
The purpose of this study is to evaluate the efficacy of Baker's yeast extractions , probiotic antioxidant, in scavenging the oxidative stress status mediated damage on sperm motility,progressive motility and vitality as well as comparing this potency to that of Vitamin E in infertile men.

DETAILED DESCRIPTION:
The practical part of the study took place from August 2020 to November 2021. The Study population was made up of infertile males attending Hawaa fertility center, banha city, Qaliubiya, Egypt.

40 study samples were collected from patients who indicated willingness to participate in the study and have had 3 to 7 days of sexual abstinence, using the masturbation method and ejaculated in wide mouthed plastic container as described by World Health Organization (WHO).

Samples were allowed to liquefy for 20 minutes and were examined for volume, viscosity, spermatozoa count by Neubauer haemocytometer , oxidative stress level measurement by Oxisperm, percentage of progressive motility and non-progressive motility and sperm vitality.

The Semen specimens were divided into ten equal fractions. First fraction was control, 0.1ml of liquefied semen mixed with 0.1ml Ham's F10 medium and incubated at 37o C for 30 minutes., 2nd: Vit. E, 3rd (Yeast extraction ( YE).Vitamin C was obtained from (Sigma, Germany), 3rd, 4th, 5th fractions (Vit. C. 1,2,3), 0.1ml liquefied semen was mixed with 0.1ml Ham's F10 medium supplemented with (0.02, 0.04, 0.06 mg/ml) Vitamin C respectively and incubated at 37o C for 30 minutes.

After semen specimen treated in all fractions, they were examined and assessed for microscopical changes, total motility, progressive motility, vitality, level of oxidative stress (OS) were detected in all fractions 30 minutes later after addition of the antioxidants.

ELIGIBILITY:
Inclusion Criteria:

* must have been married for 1 year before inclusion into the study and were unable to achieve pregnancy
* must have not received an antibiotic treatment for the last 4 weeks prior to sampling
* showed oxidative stress- mediated asthenozoospermia in their semen

Exclusion Criteria:

* Severe male Factor

Ages: 22 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
total motile sperm | 30 minutes
  Number of motile sperms in prepared semen sample per high power field (HPF)
progressive motile sperm | 30 minutes
  Number of progressively-motile sperms in prepared semen sample per HPF
vitality | 30 minutes
  Number of Vital sperms in prepared semen sample per HPF
oxidative stress | 30 minutes
  level of oxidative stress (OS) By Oxisperm Kit

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S Saad, MD, Principal Investigator — Benha University
Locations (1):
- hawaa Fertility center, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
not decided yet, but the data will be shared